CLINICAL TRIAL: NCT01048567
Title: Use of Lactobacillus Acidophilus/Rhamnosus Complex for the Prevention of Antibiotic-associated Diarrhea in Elderly Hospitalized Patients
Brief Title: Efficacy and Safety of Lactobacillus Acidophilus/Rhamnosus Combination for the Prevention of Antibiotic-associated Diarrhea in the Elderly
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient resources to meet enrollment target
Sponsor: Vancouver Island Health Authority (Other)
Collaborators: Jamieson Laboratories Ltd, Canada (Unknown); Canadian Society of Hospital Pharmacists (Other)
Responsible Party: Principal Investigator, Curtis Harder, Clinical Pharmacy Specialist, Vancouver Island Health Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIHA2009-82
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Diarrhea; Clostridium Difficile
Keywords: Antibiotics; Diarrhea; Clostridium difficile; Probiotics; Prevention & control
MeSH Terms: conditions — Diarrhea | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus acidophilus/rhamnosus (Active Comparator)
  Interventions: Other: Lactobacillus acidophilus/rhamnosus
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lactobacillus acidophilus/rhamnosus — 2 capsules (at least 2 billion cells per capsule) three times daily for duration of antibiotic therapy
  Other Names: Lactobacillus Acidophilus Probiotic Complex (by Jamieson Laboratories Ltd, Canada)
  Arms: Lactobacillus acidophilus/rhamnosus
Other: Placebo — 2 capsules three times daily for entire duration of antibiotic therapy.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Lactobacillus acidophilus/rhamnosus complex is effective in the prevention of antibiotic-associated diarrhea (AAD) in the elderly.

DETAILED DESCRIPTION:
Antibiotic-associated diarrhea (AAD) is a common adverse drug reaction, occurring in 5-35% of patients, and is of significant consequence to hospitalized patients. Patients who develop AAD are more likely to experience a longer hospital stay, incur higher medical costs, and develop other co-morbidities. Clostridium difficile infection (CDI) accounts for approximately 15-25% of AAD cases and is a significant cause of morbidity and mortality in hospitalized geriatric patients.

A preventative measure that has been suggested for AAD and CDI is the use of probiotics. Although probiotics have been used for a wide range of indications, including the prevention and treatment of AAD and CDI, there is lack of data regarding efficacy of these products.

Hospitalized elderly patients are at significant risk of developing AAD and CDI and prevention of AAD and CDI in this population may contribute to a reduction in morbidity, length of hospital stay, medical costs, and potentially mortality.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients over the age of 60 on 4A/B unit at Victoria General Hospital, Victoria BC, and
* Anticipated to receive antibiotics (intravenous or oral) for greater than 72 hours for any indication, and
* Are determined to be competent by the prescriber.

Exclusion Criteria:

* Patients who have been on antibiotics during the past 2 weeks
* Patients who have active diarrhea at enrollment
* Patients who have been diagnosed with CDI within the previous 3 months
* Patients who are lactose intolerant
* Patients who have an underlying chronic GI tract disease (inflammatory bowel disease, irritable bowel syndrome)
* Patients who have an ileostomy or colostomy
* Patients who regularly take probiotics
* Patients who are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year)
* Patients who have a life-threatening illness
* Patients who cannot take medications by mouth or are tube fed
* Patients who have been on the new antibiotic for more than 72 hours
* Patients who are anticipated to receive the new antibiotic for a duration of less than 72 hours
* Patients who do no give informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of AAD defined as 3 or more loose stools in a 24 hour period. | Monitored cnce daily at start of study product, then weekly x 3 weeks after last antibiotic dose

SECONDARY OUTCOMES:
Incidence of CDI as detected by a stool assay (detection of toxins A or B) | Measured if diarrhea develops in hospital during antibiotic treatment or during the 3 weeks following last antibiotic dose
Duration of hospital stay | Day of hospital admission until day of discharge
Incidence of adverse effects | Monitored daily at start of study product, then weekly x 3 weeks after last antibiotic dose

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Harder, BSc. Pharm, ACPR, Pharm D, Principal Investigator — Vancouver Island Health Authority
Locations (1):
- General Medicine Unit 4 A/B at Victoria General Hospital, Vancouver Island Health Authority, Victoria, British Columbia, Canada